CLINICAL TRIAL: NCT01021501
Title: the Effect of Nifedipine Controlled Release Tablets in Hypertensive Patients on Chronic Maintenance Hemodialysis and the Influence of Hemodialysis on the Plasma Concentration of Nifedipine
Brief Title: The Pharmacokinetics of Nifedipine Controlled Release Tablets in Hypertensive Patients on Hemodialysis
Acronym: PICASSO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Junzhou Fu, Nephrology department of Guangzhou First Municipal People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: GZSYIC002
Record Dates: First submitted 2009-11-27; First posted 2009-11-30 (Estimated); Last update posted 2009-11-30 (Estimated); Status verified 2009-11

CONDITIONS: Hypertension on Chronic Maintenance Hemodialysis
Keywords: nifedipine controlled release tablets; hypertensive; chronic maintenance hemodialysis; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nifedipine controlled release tablets (Experimental): Prospective, open, non-randomized, non-controlled study to evaluate the effect and safety of nifedipine controlled release tablets in hypertensive patients on chronic maintenance hemodialysis and the influence of hemodialysis on the plasma concentration of nifedipine
  Interventions: Drug: nifedipine controlled release tablets

INTERVENTIONS:
Drug: nifedipine controlled release tablets — nifedipine controlled release tablets 60mg/day for at least 4 weeks
  Other Names: Adalat GITS

SUMMARY:
This is a prospective, open, non-randomized, non-controlled study. 20 patients with hypertension on chronic maintenance hemodialysis will be enrolled in the study. All patients had mild to moderate hypertension and are receiving antihypertensive agents.

This study was designed to investigate effects of Adalat GITS on hemodialytic blood pressures in patients with chronic hemodialysis by using ABPM and measuring the drug plasma concentrations. For the purpose of investigating the influence of hemodialysis on the drug plasma concentration as well as its efficacy, it should be necessary to assign the subjects with the Adalat monotherapy. Since most patients in the hemodialysis center will be those who need and already receive combination therapy, it would be practical to start Adalat 60mg/day monotherapy to remain similar antihypertensive effect when discontinuing the previous treatment in this study population to be screened and enrolled. And taking into the consideration of clinical practice, few patients undergoing hemodialysis could be well controlled by low dose Adalat 30mg/day alone. So this study will evaluate the effect and safety of Adalat GITS 60mg/day alone and thereafter the influence of hemodialysis on the drug plasma concentration without any other possible drug interaction. The agents are given orally once a day at 08:00h and patients are followed for at least 4 weeks. After that,the patients whose blood pressure are well controlled by Adalat GITS 60mg/day by office blood pressure would be enrolled for further ABPM assessment and plasma concentration evaluation.

DETAILED DESCRIPTION:
Calcium channel blockers are widely used to reduce blood pressure in hypertensive patients on hemodialysis. They are useful I patients with left ventricular hypertrophy, diastolic dysfunction and stable angina pectoris. Adalat GITS, a long-acting dihydropyridine calcium channel blocker, has been used as one of first choices to treat the hypertension because of its effective hypotensive potency and relative absence of side effects compared with the short-acting agent. Antihypertensive effects of calcium channel blockers largely depend on their plasma concentrations, a rapid increase in blood pressure may occur as circulating levels of such blockers decrease after hemodialysis. This rapid fluctuation in blood pressure may evoke rapid alteration in hemodynamics. Luik et al. show that pre- or post-dialysis blood pressure measurements in patients with hemodialysis may be misleading for determining the blood pressure. Ambulatory pressure monitoring (ABPM) may be more useful for estimating blood pressure control in the dialysed patients. For most patients on dialysis, the goal office blood pressure is less than an average value below 150/90 mmHg on no medication. The reasonable target goal of mean ambulatory blood pressure is less than 135/85 mmHg during the day and less than 120/80 mmHg at night.

There is need of more convincing data to demonstrate the effect of Adalat GITS on hemodialytic patients by using ABPM and investigating the plasma concentrations. This study was designed to investigate effects of Adalat GITS on hemodialytic blood pressures in patients with chronic hemodialysis by using ABPM and measuring the drug plasma concentrations.

This is a prospective, open, non-randomized, non-controlled study. 20 patients with hypertension on chronic maintenance hemodialysis will be enrolled in the study. All patients had mild to moderate hypertension and are receiving antihypertensive agents.

All antihypertensive agents received by patients screened were withdrawn and patients are assigned to receive only nifedipine controlled release tablets 60mg/day. The agents are given orally once a day at 08:00h and patients are followed for at least 4 weeks. After 4 weeks of antihypertensive treatment, 20 patients with adequate blood pressure achieved (pre-hemodialysis office blood pressure < 140/90 mmHg) will be recruited into the study. If adequate blood pressure is not achieved, the patients will be excluded.

After patients have achieved adequate blood pressure (pre-hemodialysis office blood pressure < 140/90 mmHg) at enrollment, 24-hour ambulatory blood pressure monitoring (ABPM) is immediately performed on the day of hemodialysis within the subsequent two days. The administration of Adalat will continue as previously until the morning of the hemodialytic day with AMPM and blood samplings for study. The blood was sampled just before, 1 hour after, 2 hour after and 3 hour after the start of hemodialysis, and immediately after hemodialysis to measure circulating levels of nifedipine and the corresponding time points on the next hemodialysis-free day.

The 24-hour ABPM is performed in each enrolled patient on the day of hemodialysis. The monitoring is started at 08:00 h when the drugs are given. The device is programmed to measure blood pressure every 30 min (from 08:00 h to 21:00 h) and every 60 min (from 21:00 h to 08:00 h).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females >= 18 years
2. The patients are on chronic maintenance hemodialysis and dialyzed three times a week for 240 minutes.
3. The patients have mild to moderate hypertension and are receiving antihypertensive agents.
4. The dry weight of all patients is stable for at least 3 months. Dry weight is defined as the end-dialysis weight that was regularly reached without signs of dehydration or overhydration.
5. Patients who have given a written informed consent.
6. Females who are not yet in menopause should have an accepted contraception. A urine pregnancy test should be done if applicable, too.

Exclusion Criteria:

1. Patients with an interdialytic increase of greater than 5% of body weight are excluded.
2. Known hypersensitivity to nifedipine or any of the ingredients
3. Moderate to severe hepatic insufficiency (ALT/AST>2 x ULN (= Upper Limit of Normal))
4. Cardiovascular disease such as atrial fibrillation, congestive heart failure, valvular or ischemic heart disease, or stroke, or life-threatening arrhythmia
5. fluid effusion
6. inflammatory disease
7. malignancies
8. Female patients who are pregnant or lactating.
9. Other contraindications in package insert.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-12 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
To investigate the effect and safety of nifedipine controlled release tablets in patients on chronic maintenance hemodialysis by using ABPM. | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Junzhou Fu, Master, Principal Investigator — Department of Nephrology, Guangzhou First Municipal People's Hospital
Locations (1):
- Department of Nephrology, Guangzhou First Municipal People's Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Kojima M, Taniguchi M, Sato K, Ueda R, Dohi Y. Antihypertensive effects of long-acting calcium channel blockers on hemodialysis days--a randomized crossover trial between benidipine and nifedipine CR. Nephron Clin Pract. 2004;97(2):c49-53. doi: 10.1159/000078400. PMID 15218330
- [Background] Martre H, Sari R, Taburet AM, Jacobs C, Singlas E. Haemodialysis does not affect the pharmacokinetics of nifedipine. Br J Clin Pharmacol. 1985 Aug;20(2):155-8. doi: 10.1111/j.1365-2125.1985.tb05049.x. PMID 4041333